CLINICAL TRIAL: NCT03347916
Title: The Role of Gabapentin Oral Solution in Decreasing Desflurane Associated Emergence Agitation and Delirium in Children After Strabismus Surgery: A Prospective Randomized Double-blind Study
Brief Title: Gabapentin Oral Solution in Decreasing Desflurane Associated Emergence Agitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kuwait Specialized Eye Center (Other)
Responsible Party: Principal Investigator, Ahmed A. Badawy, Anesthesia Consultant, Kuwait Specialized Eye Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: kuwaiteyecenter01
Record Dates: First submitted 2017-11-14; First posted 2017-11-20 (Actual); Last update posted 2017-11-21 (Actual); Status verified 2017-11

CONDITIONS: Emergence Agitation After Desflurane Anesthesia
MeSH Terms: interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): patients received strawberry juice 5 ml volume, one hour before induction.
  Interventions: Drug: Strawberry juice as (placebo)
- Gabapentin group (Active Comparator): patients received gabapentin (Neurontin oral solution 250 mg/ml, Pfizer, USA) 5 mg/kg mixed with strawberry juice to constitute 5 ml volume, one hour before induction.
  Interventions: Drug: Gabapentin Oral Solution [Neurontin]

INTERVENTIONS:
Drug: Strawberry juice as (placebo) — Patients received strawberry juice 5 ml volume, one hour before induction.
  Other Names: Strawberry juice
  Arms: Control group
Drug: Gabapentin Oral Solution [Neurontin] — Patients received gabapentin (Neurontin oral solution 250 mg/ml, Pfizer, USA) 5 mg/kg mixed with strawberry juice to constitute 5 ml volume, one hour before induction.
  Other Names: Neurontin
  Arms: Gabapentin group

SUMMARY:
to study the effect of oral gabapentin (5 mg/kg) on emergence agitation after desflurane anesthesia in pediatrics undergoing starbismus surgery

ELIGIBILITY:
Inclusion Criteria:

* pediatric patients (2-6 years old), with an American society of Anesthegiologists physical status (ASA) I-II who were undergoing strabismus surgery (for more than one muscle)

Exclusion Criteria:

* failure to obtain consent, mental retardation or developmental delay, epilepsy, psychiatric or neurological diseases that impair communication, current use of gabapentin, psychotropic or opioids.

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Estimated)
Dates: Start 2017-01-05 (Actual); Primary Completion 2017-11-25 (Estimated); Study Completion 2017-11-30 (Estimated)

PRIMARY OUTCOMES:
emergence agitation incidence and scores | through study completion, an average of 1 year
  agitation measured by emergence agitation scale: [1= Obtunded with no response to stimuli; 2= Asleep, but responsive to movement and stimuli; 3= Awake and appropriately responsive; and 4= Crying and difficult to console; 5= Wild thrashing behaviour that requires restraint]. A score 4 or 5 was considered as agitation and was treated by IV meperidine 0.5 -1 mg/kg increments.

SECONDARY OUTCOMES:
duration of emergence | through study completion, an average of 1 year
  The time from the discontinuation of anesthesia till the time of spontaneous eye opening or to verbal command

CONTACTS AND LOCATIONS:
Locations (1):
- Kuwait Specialized Eye Center, Kuwait City, Kuwait

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Badawy AA, Kasem SA, Rashwan D, Al Menesy T, Adel G, Mokhtar AM, Badawy YA. The role of Gabapentin oral solution in decreasing desflurane associated emergence agitation and delirium in children after stabismus surgery, a prospective randomized double-blind study. BMC Anesthesiol. 2018 Jun 20;18(1):73. doi: 10.1186/s12871-018-0533-5. PMID 29925328